CLINICAL TRIAL: NCT02504801
Title: Efficacy of Nebulized Pulmicort Respules on Post Operation Pulmonary Complication During Pulmonary Single Lobectomy Surgery in Primary Lung Cancer Patients With COPD
Brief Title: Efficacy of Nebulized Pulmicort Respules in Primary Lung Cancer Patients With COPD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xiuyi Zhi (Other)
Responsible Party: Sponsor-Investigator, Xiuyi Zhi, Professor, Xuanwu Hospital, Beijing
Organization: Xuanwu Hospital, Beijing (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ISSPULR0007
Record Dates: First submitted 2015-07-15; First posted 2015-07-22 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Post Operative Complication, Pulmonary; Lung Cancer; COPD
Keywords: primary lung cancer patients
MeSH Terms: conditions — Lung Neoplasms; Pulmonary Disease, Chronic Obstructive | interventions — Budesonide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- nebulized Budesonide 2mg/4mL (Active Comparator): +terbutaline 5mg/2mL,BID+ipratropium 2 puff(40ug)BID
  Interventions: Drug: Budesonide
- nebulized saline 4mL (Placebo Comparator): +terbutaline 5mg/2mL,BID+ipratropium 2 puff(40ug)BID

INTERVENTIONS:
Drug: Budesonide — To test the hypothesis that nebulizer Pulmicort Respules could reduce post operation pulmonary complication incidence in primary lung cancer patients with COPD. Compare post-operation pulmonary complication incidence in two arms among primary lung cancer patients with COPD required single lobectomy from 3 days before operation to 7 days after operation.
  Arms: nebulized Budesonide 2mg/4mL

SUMMARY:
To test the hypothesis that nebulized Pulmicort Respules could reduce post operation pulmonary complication incidence in primary lung cancer patients with COPD. Compare post-operation pulmonary complication incidence in two treatment arms among primary lung cancer patients with COPD required single lobectomy from 3days before operation to 7 days after operation.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed or existing COPD defined by GOLD, and FEV1 of<80% predicted and FEV1/FVC<70%
2. Diagnosed as primary lung cancer by China guidelines on diagnosis and treatment of primary lung cancer
3. .Consistent with indication of operation of pulmonary single lobectomy surgery by China guidelines on diagnosis and treatment of primary lung cancer
4. General anesthesia and double cavity intubation was used during operation
5. ASA Classification of Anesthesia Risk is in category 1-3 both in baseline
6. age from 40-80 years old
7. Smoking cessation more than two weeks before operation
8. SP O2>90% before surgery
9. Hemoglobin > 10g/dl
10. Estimated duration of surgery < 4 hours
11. 18.5<BMI < 28

Exclusion Criteria:

1. Patients who had taken systemic corticosteroids in the preceding 1month before baseline
2. Patients who had pneumonia in the preceding 1month before baseline
3. Patients with a history of recent myocardial infarction, heart failure, tuberculosis
4. Subject with known or suspected human immunodeficiency virus infection

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2015-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
The incidence of post-operation pulmonary complication in two arms among primary lung cancer patients with COPD | 10 days
  Definition of post-operation pulmonary complication:
  1. Pneumonia/other pulmonary infections, with X-ray evidence, fever and/or WBC>15,000mL
  2. Sputum retention:classified as purulent and the pour ability grade is 1 or 2
  3. Acute respiratory failture or chronic respiratory failture
  4. Atelectasis
  5. Aerothorax:>30% by X-ray; pulmonary embolism